CLINICAL TRIAL: NCT07201246
Title: Retrospective Analysis of Organ Dysfunction Changes in Acute Necrotizing Pancreatitis Patients With Sepsis Following Open Necrosectomy：A Retrospective Cohort Study
Brief Title: Organ Dysfunction Changes in Acute Necrotizing Pancreatitis Patients With Sepsis Following Open Necrosectomy
Status: Not yet recruiting | Type: Observational
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Chunling Jiang, Professor, West China Hospital
Other Study IDs: 2024-162
Record Dates: First submitted 2025-09-18; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Necrotizing Pancreatitis
MeSH Terms: conditions — Pancreatitis, Acute Necrotizing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pancreatitis with sepsis patients' organdysfunction progression after opennecrosectomy: SOFA scores at predefined time points were retrospectively extracted from the institutional database in acute necrotizing pancreatitis patients with sepsis who underwent open necrosectomy to characterize organ dysfunction trajectories
  Interventions: Other: Necrotizing Pancreatitis patients' organdysfunction progression

INTERVENTIONS:
Other: Necrotizing Pancreatitis patients' organdysfunction progression — Study the dynamic nature of organ dysfunction

SUMMARY:
The purpose of this retrospective study was to characterize the changes in organ dysfunction among patients with acute necrotizing pancreatitis complicated by sepsis who underwent open necrosectomy.

DETAILED DESCRIPTION:
Baseline demographic and clinical characteristics (including age, gender, and education level) were collected from medical records. Organ dysfunction was defined according to the Sequential Organ Failure Assessment (SOFA) score. SOFA scores were extracted at predefined time points: preoperative (T1), postoperative day 1 (T2), postoperative day 3 (T3), and either postoperative day 7 or hospital discharge, whichever occurred first (T4). Postoperative survival status up to 1 year was obtained from the institutional database.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 years or older
2. Diagnosis of Acute pancreatitis according to the revised Atlanta classification, requires two of thefollowing three criteria: (A) typical abdominal pain, (B) an increase in serum amylase or lipaselevels higher than three times the upper limit of normality, and (C) signs of AP in imaging3)Patients with confirmed or suspected infected pancreatic or peripancreatic necrosis werescheduled for open necrosectomy
3. Meet Sepsis-3 criteria

Exclusion Criteria:

Patients undergo repeat surgery on the same site

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This retrospective cohort included patients with acute necrotizing pancreatitis complicated by sepsis who underwent open necrosectomy
Sampling Method: Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2025-10-05 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Measure organ dysfunction change after open necrosectomy with respect to time | up to postoperative day 7, or at hospital discharge, whichever comes first
  Organ dysfunction was assessed retrospectively using the Sequential Organ Failure Assessment (SOFA) score, which ranges from 0 (normal) to 4 (most abnormal) for each organ, with higher scores indicating more severe dysfunction.

SECONDARY OUTCOMES:
Incidence of ICU mortality | an average of 1year
Incidence of hospital mortality | an average of 1 year
Incidence of 28-day mortality | an average of 1 year
Incidence of one year mortality | an average of 1 year
ICU length of hospital stay | an average of 1 year
Length of hospital stay | an average of 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital, Sichuan University, Chengdu, China, China

IPD SHARING:
Plan to Share IPD: No